CLINICAL TRIAL: NCT02743026
Title: An Arts-based HIV and Sexually Transmitted Infection Prevention Intervention With Northern and Indigenous Youth in the Northwest Territories: Study Protocol for a Non-randomised Cohort Pilot Study
Brief Title: HIV and Sexually Transmitted Infection Prevention Intervention in the Northwest Territories
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Carmen Logie, MSW, PhD, Assistant Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIHR-CBR-0000303157
Record Dates: First submitted 2016-04-11; First posted 2016-04-19 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: HIV; Sexually Transmitted Diseases
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — 6-fluoro-6-desoxyoxymorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): participants will complete the FOXY intervention
  Interventions: Behavioral: FOXY

INTERVENTIONS:
Behavioral: FOXY — This study will evaluate an arts-based HIV prevention program, Fostering Open eXpression among Youth (FOXY) in the NWT, Canada that works with Northern and Indigenous youth to promote sexual health and reduce exposure to HIV/STI. FOXY explores sexual health, HIV/STIs, sexuality and healthy relationships with young women in the NWT. The program's goal is to use arts-based methods and peers to facilitate education and foster more open expression and communication regarding sexual health and sexuality. FOXY uses arts-based approaches in program delivery; for example, drama techniques are used to facilitate discussion and learning about healthy relationships and making positive choices in realistic sexual scenarios.

SUMMARY:
Indigenous youth are disproportionately represented in new HIV infection rates in Canada. Limited studies have evaluated longitudinal effects of arts-based approaches to HIV prevention with youth. The authors present a rationale and study protocol for an arts-based HIV and sexually transmitted infections (STI) prevention intervention with Northern and Indigenous youth in the Northwest Territories (NWT), Canada. This is a multi-centre non-randomised cohort pilot study using a pre-test/post-test design with a 12-month follow-up. The target population is Northern and Indigenous youth in eighteen communities in the NWT. The aim is to recruit 150 youth using venue-based sampling at secondary schools. Participants will be involved in an arts-based intervention, Fostering Open eXpression among Youth (FOXY). Participants will complete a pre-test, post-test survey directly following the intervention, and a 12-month follow up.

DETAILED DESCRIPTION:
Introduction: Indigenous youth are disproportionately represented in new HIV infection rates in Canada. Current and historical contexts of colonization and racism, disconnection from culture and land, as well as intergenerational trauma resulting from the legacy of residential schools are social drivers that elevate exposure to HIV among Indigenous peoples. Peer-education and arts-based interventions are increasingly used for HIV prevention with youth. Yet limited studies have evaluated longitudinal effects of arts-based approaches to HIV prevention with youth. The authors present a rationale and study protocol for an arts-based HIV prevention intervention with Northern and Indigenous youth in the Northwest Territories (NWT), Canada.

Methods & Analysis: This is a multi-centre non-randomised cohort pilot study using a pre-test/post-test design with a 12-month follow-up. The target population is Northern and Indigenous youth in eighteen communities in the NWT. The aim is to recruit 150 youth using venue-based sampling at secondary schools. Participants will be involved in an arts-based intervention, Fostering Open eXpression among Youth (FOXY). Participants will complete a pre-test, post-test survey directly following the intervention, and a 12-month follow up. The primary outcome is new or enhanced HIV knowledge, and secondary outcomes to include: new or enhanced STI knowledge, and increased self-esteem, resilience, empowerment, safer sex self-efficacy, and cultural connectedness. Mixed effects regression analyses will be conducted to evaluate pre- and post-test differences in outcome measurement scores.

Ethics and Dissemination: This study has received approval from the HIV Research Ethics Board at the University of Toronto (REB: 31602).

ELIGIBILITY:
Inclusion Criteria:

* participating in FOXY
* self-identify as a woman
* live in the Northwest Territories
* between the ages of 13 and 16 years of age
* capable of providing informed consent

Exclusion Criteria:

* did not participate in FOXY
* not between 13-16 years old
* don't live in the Northwest Territories
* not capable of providing informed consent

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 199 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
HIV knowledge (Questionnaire) | 12 month follow up
  Brief HIV Knowledge Questionnaire

SECONDARY OUTCOMES:
Sexually Transmitted Infections knowledge (Questionnaire) | 12 month follow up
  Sexually Transmitted Disease Knowledge Questionnaire
Self-esteem (scale) | 12 month follow up
  Self-esteem scale
safer sex self-efficacy (Scale) | 12 month follow up
  Safer Sex Self-Efficacy Scale
cultural connectedness (Scale) | 12 month follow up
  Awareness of Connectedness Scale

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Logie, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Factor-Inwentash Faculty of Social Work, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Small numbers in towns in the North make it difficult to share data without compromising confidentiality.

REFERENCES:
- [Background] Lys C, Reading C. Coming of age: how young women in the Northwest Territories understand the barriers and facilitators to positive, empowered, and safer sexual health. Int J Circumpolar Health. 2012 Jul 2;71:18957. doi: 10.3402/ijch.v71i0.18957. PMID 22765935
- [Derived] Lys C, Logie CH, MacNeill N, Loppie C, Dias LV, Masching R, Gesink D. Arts-based HIV and STI prevention intervention with Northern and Indigenous youth in the Northwest Territories: study protocol for a non-randomised cohort pilot study. BMJ Open. 2016 Oct 3;6(10):e012399. doi: 10.1136/bmjopen-2016-012399. PMID 27697877